# WRITTEN INFORMED CONSENT

# INFORMED CONSENT FORM COVER PAGE

#### **Official Study Title**

Behavioral Interventions for Multiple Micronutrient Supplement Adherence in Cambodian Pregnancy: A Mixed-Methods Study

## **Study Information**

- NCT Number: To be assigned by ClinicalTrials.gov
- Document Date: September 22, 2024
- Document Type: Written Informed Consent

# Informed Consent Form for Research Study on Nutrition Supplementation during Pregnancy

#### 1. Introduction

My name is [Your Name], and I am from Helen Keller International (HKI) Cambodia. Helen Keller Intl is a non-profit organization working on health, nutrition, and agriculture. We are collaborating with the Ministry of Health in Cambodia to research pregnant women's experiences with interventions and strategies to help them take prenatal supplements.

#### 2. Purpose of the Study

This study aims to understand what strategies and social support can improve women's acceptance and adherence to nutrition supplements in Cambodia. The information we gather will help enhance programs and policies for nutrition supplementation during pregnancy, ultimately aiming to benefit the health of mothers and babies in Cambodia.

#### 3. Why You Are Being Asked to Participate

You are being invited to participate because you are pregnant and enrolled in antenatal care visits at a health facility involved in the study. Your participation will be valuable as it provides insights from pregnant women receiving these supplements.

#### 4. Procedures

We are encouraging you to take a safe and effective nutrition supplement as part of your regular antenatal care. We would like to understand your experience with these supplements, including how often you take them, any side effects you experience, and any concerns you may have.

We will also invite some members of your household to attend a 30-minute orientation session to provide them with information on the importance of prenatal supplementation during pregnancy and how to support you during this time. After one month, you will receive a wall calendar to put up in your home. The calendar will provide information on how to have a healthy pregnancy.

We may invite you to attend three focus group discussions each month to discuss your experiences with the nutrition supplements you receive during your ANC visits.

#### 5. Risks and Discomforts

There is no physical risk associated with this study. You may experience some discomfort answering personal questions. You are free to skip any questions you feel uncomfortable with.

#### 6. Benefits

There is no direct benefit to you for participating in this study. However, your participation will improve pregnant women's and babies' health and well-being in Cambodia by informing better nutrition supplementation programs.

#### 7. Protecting Data Confidentiality

All your information will be kept strictly confidential. Your name will not be used in any reports or publications from this study. We will assign a code number to your data to protect your privacy.

#### 8. Payment

There is no financial compensation for participating in this study, but you will be given a small token gift each time you participate in the focus group discussion, and you will be given a wall calendar that gives you information on what to expect during pregnancy and information on how to stay healthy during your pregnancy.

## 9. Voluntary Participation

Your participation in this study is entirely voluntary. You can withdraw your consent and discontinue participation at any time without penalty.

#### 10. Questions and Concerns

If you have any questions or concerns about the study, please do not hesitate to ask me or contact:

Meng Sokchea (Project Manager, HKI Cambodia)

Email: msokchea@hki.org Mobile: 012 61 2 912

#### 11. Your Decision

Thank you for considering participating in this study. Please take your time to decide; there is no pressure to participate.

If you agree to participate, please sign below.

| Name of person giving consent: |
|---|
| Signature of person giving consent: |
| Date of obtained consent: |
| Name of research staff obtaining consent: |
| I give HKI permission to take photos or videos of me for any purpose with the |